CLINICAL TRIAL: NCT03931291
Title: Phase II Trial of APR-246 in Combination With Azacitidine as Maintenance Therapy for TP53 Mutated AML or MDS Following Allogeneic Stem Cell Transplant
Brief Title: APR-246 in Combination With Azacitidine for TP53 Mutated AML (Acute Myeloid Leukemia) or MDS (Myelodysplastic Syndromes) Following Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A19-11172
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia or Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — eprenetapopt; Azacitidine

STUDY DESIGN:
Intervention Model Description: APR-246 will be administered on Days 1-4, with azacitidine on Days 1-5, of every 28 day cycle. Patients may receive a maximum of 12 cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental arm: APR-246 + azacitidine (Experimental): APR-246 and azacitidine maintenance therapy will continue for a maximum of 12 cycles
  Interventions: Drug: APR-246

INTERVENTIONS:
Drug: APR-246 — APR-246 will be administered on Days 1-4, with azacitidine on Days 1-5, of every 28 day cycle. Patients may receive a maximum of 12 cycles.
  Other Names: Azacitidine

SUMMARY:
A multi-center, open label, Phase II clinical trial to assess the safety and efficacy of APR-246 in combination with azacitidine as maintenance therapy after allogeneic HSCT (hematopoietic stem cell transplant) for patients with TP53 mutant AML or MDS.

DETAILED DESCRIPTION:
A multi-center, open label, Phase II clinical trial to assess the safety and efficacy of APR-246 in combination with azacitidine as maintenance therapy after allogeneic HSCT for patients with TP53 mutant AML or MDS.

Patients will be prescreened for TP53 mutant AML or MDS before they have a HSCT. In order to proceed with APR-246 and azacitidine treatment, engraftment must be confirmed between Day 30 to Day 100 post-HSCT.

APR-246 will be administered on Days 1-4, with azacitidine on Days 1-5, of every 28 day cycle. Patients may receive a maximum of 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have previously met pre-transplantation eligibility.
2. Patient has received an allogeneic transplant for AML or MDS.
3. Any standard (non-study) conditioning [MAC (myeloablative conditioning), RIC (reduced intensity conditioning), or NMA (non-myeloablative conditioning)] will be permitted.
4. Patient is ≥ 30 days and ≤ 100 days from hematopoietic cell infusion.
5. Patient is in complete remission after the transplant and has achieved engraftment. .
6. Patients who have developed grades II-IV acute GVHD (graft versus host disease) will be allowed to initiate maintenance therapy based on the following criteria:
7. Females must either:

   Be of non-childbearing potential postmenopausal (defined as at least 1 year without menses) prior to screening, or documented as surgically sterilized (e.g., hysterectomy or tubal ligation) at least 1 month prior to the screening visit Or, if of childbearing potential, Agree not to try to become pregnant during the study and for 6 months after the final study drug administration And have a negative serum pregnancy test at screening And, if heterosexually active, agree to consistently use highly effective contraception per locally accepted standards in addition to a barrier method starting at screening and throughout the study period and for 6 months after final study drug administration.
8. Females must agree not to breastfeed or donate ova throughout the study drug treatment period and for 6 months after the final study drug administration.
9. Males (even if surgically sterilized), and their partners who are women of childbearing potential must be using highly effective contraception in addition to a barrier method throughout the study drug treatment period.
10. Males must not donate sperm throughout the study drug treatment period.
11. Agrees not to participate in another interventional study while on treatment.
12. Karnofsky Performance Status 70 or greater is required.

Exclusion Criteria:

1. Prior participation in an APR-246 study.
2. Use of umbilical cord blood donor and stem cell source.
3. Patient has uncontrolled infection.
4. Use of investigational agent within 14 days of pre-HSCT screening or anytime thereafter.
5. Use of hypomethylating agent, cytotoxic chemotherapeutic agents, or experimental agents (agents that are not commercially available) for the treatment of MDS or AML within 14 days of the first day of pre-HSCT screening or anytime thereafter.
6. Patient has used experimental therapy for acute GVHD at any time post-transplant.
7. Patient requires treatment with supplemental oxygen not including usage of non-invasive CPAP (continuous positive airways pressure) at night.
8. Patient has any of the following cardiac abnormalities (as determined by treating physician):

   1. Myocardial infarct within six months prior to registration
   2. New York Heart Association Class II or worse heart failure or known LVEF (left ventricular ejection fraction) < the institution LLN (lower limit normal)
   3. A history of familial long QT syndrome
   4. Electrocardiographic evidence of acute ischemia at screening
   5. Symptomatic atrial or ventricular arrhythmias not controlled by medications
   6. QTc ≥ 470 ms calculated from a mean of 3 ECG (electrocardiogram) readings using Fridericia's correction (QTcF = QT/RR0.33)
   7. Bradycardia (<40 bpm) at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asmita Mishra, MD, PhD, Principal Investigator — H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida 33612
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Johns Hopkins, Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Mishra A, Tamari R, DeZern AE, Byrne MT, Gooptu M, Chen YB, Deeg HJ, Sallman D, Gallacher P, Wennborg A, Hickman DK, Attar EC, Fernandez HF. Eprenetapopt Plus Azacitidine After Allogeneic Hematopoietic Stem-Cell Transplantation for TP53-Mutant Acute Myeloid Leukemia and Myelodysplastic Syndromes. J Clin Oncol. 2022 Dec 1;40(34):3985-3993. doi: 10.1200/JCO.22.00181. Epub 2022 Jul 11. PMID 35816664

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm: APR-246 + Azacitidine
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm: APR-246 + Azacitidine
Number analyzed (Participants) | 33
Age, Customized [Median (Full Range); unit: years] | 65 [40 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: To Assess Relapse-free Survival (RFS) in Patients With TP53 Mutated AML or MDS After Undergoing Allogeneic Hematopoietic Stem Cell Transplant (HSCT).
Description: Relapse-free survival (RFS) at 12 months or longer if data permits. RFS was defined as the time from HCT to relapse after HCT or death, whichever occurred first.
Time Frame: Through study completion, an average of 1 year
Population: Allogenic Transplant Patients with TP53 AML or MDS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm: APR-246 + Azacitidine
Number analyzed (Participants) | 33
months | 12.5 [9.6 to 14.5]

ADVERSE EVENTS:
Time Frame: 13 months
Description: The AE reporting period starts from the day of signing the post-transplant informed consent form. AEs will be collected for 30 days after the last dose of study drug.
Arm/Group | Experimental Arm: APR-246 + Azacitidine
All-Cause Mortality (participants affected / at risk) | 13/33
Serious Adverse Events (participants affected / at risk) | 13/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: APR-246 + Azacitidine (N=33)
Pyrexia (General disorders) | 4
Disease progression (General disorders) | 1
General Oedema (General disorders) | 1
Malise (General disorders) | 1
Pain (General disorders) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 3
Seroma (Injury, poisoning and procedural complications) | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Device related infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viremia (Infections and infestations) | 1
Blood Bilirubin Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Dysponea (Respiratory, thoracic and mediastinal disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain Lower (Gastrointestinal disorders) | 1
Confusional state (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: APR-246 + Azacitidine (N=33)
Nausea (Gastrointestinal disorders) | 20
Platelet Count Decreased (Investigations) | 16
Vomitting (Gastrointestinal disorders) | 15
Anemia (Blood and lymphatic system disorders) | 13
Dizziness (Nervous system disorders) | 13
White blood cell count decreased (Investigations) | 13
Fatigue (General disorders) | 12
Diarrhea (Gastrointestinal disorders) | 11
Tremor (Nervous system disorders) | 11
Neutrophil Count decreased (Investigations) | 9
cough (Respiratory, thoracic and mediastinal disorders) | 8
pruritus (Skin and subcutaneous tissue disorders) | 8
Pyrexia (General disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 7
Consitpation (Gastrointestinal disorders) | 7
Decreased Appetite (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 7
Dry Mouth (Gastrointestinal disorders) | 6
Dyskinesia (Nervous system disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypertension (Vascular disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Blood cholesterol Increased (Investigations) | 5
Blood Creatinine Increased (Investigations) | 5
Dry Eye (Eye disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Dysuria (Renal and urinary disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 5
Insomnia (Psychiatric disorders) | 5
Edema Peripheral (General disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Ataxia (Nervous system disorders) | 4
Blood Alkaline Phosphate Increased (Investigations) | 4
Blood Lactate Dehydrogenase Increased (Investigations) | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Serum ferritin increased (Investigations) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03931291/Prot_SAP_000.pdf